CLINICAL TRIAL: NCT01561807
Title: A Phase 2a, Randomized, Double-Blind,Placebo-Controlled Study to Investigate the Effects of VX-787 Administered to Adult Volunteers Experimentally Inoculated With Live Influenza Virus
Brief Title: A Study to Investigate VX-787 Given to Adult Volunteers Inoculated With Live Influenza Virus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VX11-787-101
Record Dates: First submitted 2012-03-19; First posted 2012-03-23 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Influenza Virus
MeSH Terms: interventions — pimodivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 787 low dose (Experimental): VX-787 low dose capsule, taken orally for 5 days
  Interventions: Drug: VX-787
- 787 high dose (Experimental): VX-787 high dose capsule, taken orally for 5 days
  Interventions: Drug: VX-787
- Placebo low dose (Experimental): Matching placebo low dose capsule, taken orally for 5 days
  Interventions: Drug: Placebo
- Placebo high dose (Experimental): Matching placebo high dose capsule, taken orally for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-787
  Arms: 787 high dose; 787 low dose
Drug: Placebo
  Arms: Placebo high dose; Placebo low dose

SUMMARY:
The purpose of this study is to determine the antiviral activity and safety of VX-787 given to healthy adult volunteers that have been inoculated with the influenza virus.

ELIGIBILITY:
Inclusion Criteria:

* Negative human immunodeficiency virus (HIV), hepatitis B (HBV) and hepatitis C(HCV) antibody screen
* Have not been vaccinated for influenza virus since 2006 or had a known influenza-like illness in the current season (as determined in the medical history), defined as in the last 12 months before Screening

Exclusion Criteria:

* Subjects who are pregnant or nursing, or who are male and have a female partner who is pregnant, nursing, or is planning to become pregnant during the study period (from at least 14 days before the first dose until 90 days of the last dose of study drug)
* Presence of any significant acute or chronic, uncontrolled medical or psychiatric illness
* Abnormal pulmonary function as evidenced by clinically significant abnormalities in spirometry
* Health care workers (including doctors, nurses, medical students and allied healthcare professionals) anticipated to have patient contact within two weeks of viral inoculation
* Intending to travel(to countries for which vaccinations are recommended or where high risk of infections exists)
* Subjects with a history of asthma, COPD, pulmonary hypertension, reactive airway disease, or any chronic lung condition of any etiology; any history during adulthood of asthma of any etiology, COPD, or any use of a bronchodilator or other asthma medication during adulthood
* Regular daily smokers
* History or evidence of autoimmune disease or known impaired immune responsiveness
* History of heart failure or any other severe cardiac abnormality including clinically significant arrhythmia
* Receipt of any investigational drug within 3 months, or prior participation in a clinical trial of any influenza vaccine, medication, or experimental respiratory viral challenge delivered directly to the respiratory tract within 1 year before viral inoculation
* Previous exposure to study drug or similar substance(s)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is viral AUC as calculated in cell culture of nasal swabs (quantitation of nasal swabs for viral infectivity by cell culture), from initiation of VX-787 treatment | up to 11 days

SECONDARY OUTCOMES:
Safety and tolerability based on assessment of adverse events, clinical laboratory assessments, 12-lead electrocardiograms (ECGs), and vital signs. | up to 33 days
Total tissue count and total mucus weight after viral inoculation | up to 10 days
Sequence analysis of the relevant target region of influenza | up to 8 days
Pharmacokinetic (PK) parameters of VX-787 | 8 days
  As measured by AUC, Cmax, tmax
Composite symptom score AUC | up to 8 days
Viral AUC calculated by RT-PCR of nasal swabs, from initiation of VX-787 treatment | up to 8 days
Duration of viral shedding by cell culture and/or RT-PCR | up to 8 days
Peak viral shedding titer by cell culture and/or RT-PCR | up to 8 days
Time to resolution from peak viral shedding by cell culture and/or RT-PCR | up to 8 days
Time to peak of composite sympton score, duration, and time to resolution of composite score from peak | up to 8 days
Peak severity of symptoms after viral inoculation | up to 8 days
Duration of influenza-like illness after viral inoculation | up to 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Jose Trevejo, MD, PhD, Study Director — Vertex Pharmaceuticals Incorporated
Locations (1):
- London, United Kingdom